CLINICAL TRIAL: NCT07227740
Title: Testosterone Deficiency and Endothelial Dysfunction in Spinal Cord Injury Related Cardiovascular Disease Mechanistic Insights and Therapeutic Prospects
Brief Title: Testosterone Deficiency and Endothelial Dysfunction After Spinal Cord Injury
Status: Recruiting | Type: Observational
Sponsor: Craig Hospital (Other)
Collaborators: University of Colorado, Boulder (Other); Denver Health and Hospital Authority (Other); University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 2301643; CDMRP-SC240119 (Other Grant/Funding Number: Congressionally Directed Medical Research Programs (CDMRP))
Record Dates: First submitted 2025-11-11; First posted 2025-11-13 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Spinal Cord Injuries; Endothelial Dysfunction; Testosterone Deficiency
Keywords: spinal cord injury; endothelial dysfunction; testosterone deficiency; extracellular vesicles; microvesicles; vasodilation; fibrinolysis
MeSH Terms: conditions — Spinal Cord Injuries; Aneurysm | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum, plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Adult Male with Subacute Traumatic Spinal Cord Injury with Normal Testosterone: 24 male participants of all races and ethnic backgrounds aged 18-89 years with a history of spinal cord injury and diagnosed with normal testosterone
  Interventions: Diagnostic Test: Intra-arterial Infusion of Vasoactive Agents; Diagnostic Test: Intra-arterial Vitamin C Infusion; Diagnostic Test: Blood Sampling
- Adult Male with Subacute Traumatic Spinal Cord Injury with Low Testosterone: 24 male participants of all races and ethnic backgrounds aged 18-89 years with a history of spinal cord injury and diagnosed with low testosterone
  Interventions: Diagnostic Test: Intra-arterial Infusion of Vasoactive Agents; Diagnostic Test: Intra-arterial Vitamin C Infusion; Diagnostic Test: Blood Sampling

INTERVENTIONS:
Diagnostic Test: Intra-arterial Infusion of Vasoactive Agents — A catheter is placed in the brachial artery of the non-dominant arm, and small doses of vasoactive drugs acetylcholine, isoproterenol, sodium nitroprusside are infused. Forearm blood flow will be measured using venous occlusion plethysmography. The purpose of this procedure is to assess endothelium-dependent and independent vasodilation by stimulating different vascular pathways. The acetylcholine infusion is to test muscarinic receptor, nitro oxide dependent, endothelium-dependent vasodilation. Isoproterenol was selected to stimulate tissue plasminogen activator based on its specificity and effectiveness at eliciting local and rapid tissue plasminogen activator release in adult humans. Sodium nitroprusside infusion is to assess endothelium-independent vasodilation.
Diagnostic Test: Intra-arterial Vitamin C Infusion — Vitamin C, a potent antioxidant, will be infused into the forearm and forearm blood flow will be re-evaluated to determine whether oxidative stress contributes to endothelial dysfunction.
Diagnostic Test: Blood Sampling — Blood will be sampled from the antecubital vein (~50 mL) for biomarker analysis. This is to assess circulating biochemical and molecular indicators of vascular health and inflammation including levels of endothelial cell derived microvesicles.

SUMMARY:
Heart attacks and strokes are among the most common causes of premature death in individuals living with spinal cord injury (SCI) and appear to occur earlier in life. The factors that lead to the heighten and accelerated risk of heart attacks and strokes in adults living with SCI remain poorly understood. The investigators aim to uncover why this happens and find ways to prevent it. Our research focuses on how important cells which line blood vessels, called endothelial cells, function after SCI. The investigators test endothelial function in live conscious people with SCI. The investigators also study signaling molecules endothelial cells release called endothelial cell derived microvesicles (EMVs), which the investigators can measure in blood to tell us the health of endothelial cells. By using these rigorous tests of vascular function, the investigators have determined that endothelial cells appear dysfunctional after SCI. The investigators also know that many men with SCI have low testosterone levels. Our team has studied testosterone's effects on endothelial dysfunction and believe low testosterone may be contributing to endothelial dysfunction after SCI. By understanding these mechanisms, the investigators hope to improve the lives of those living with SCI and reduce their risk for heart attacks and strokes. The investigators propose to study the influence of testosterone on endothelial function by using state-of-the-art clinical and laboratory experiments to assess endothelial function in men with SCI with low and normal testosterone levels.

DETAILED DESCRIPTION:
The vascular endothelium plays a central role in atherosclerotic cardiovascular disease and may contribute to the increased risk of myocardial infarction and stroke following spinal cord injury (SCI). Endothelial dysfunction is characterized by impaired vasodilator function and reduced fibrinolytic capacity.

Endothelium-dependent vasodilation is primarily mediated by nitric oxide (NO), which induces rapid relaxation of vascular smooth muscle. Fibrinolysis is the breakdown of thrombi within blood vessels, and is facilitated by endothelial cells through the synthesis and release of tissue-type plasminogen activator (t-PA). Importantly, endothelial dysfunction often precedes detectable atherosclerosis and predicts future major vascular events.

Low testosterone (T) is a common secondary complication that occurs early after SCI, with hypogonadism being four times more prevalent in men with SCI. Testosterone has known antioxidant properties and its deficiency may contribute to endothelial dysfunction. Testosterone deficiency may represent a modifiable risk factor for vascular impairment after SCI.

This cross-sectional study will include 48 adults with subacute (<6 months), motor-complete (AIS A/B) paraplegia (neurological level T3 or below). 24 with testosterone deficiency and 24 with normal T levels. Endothelium-dependent vasodilation and t-PA capacity will be assessed via intra-arterial infusion of vasoactive drugs, with total forearm blood flow measured using venous occlusion plethysmography.

ELIGIBILITY:
Inclusion Criteria:

* Between ages 18-89 years of age
* Male Sex
* History of motor complete (AIS A/B) paraplegia (NLI T3 or Below)
* Time since injury <6 months at time of enrollment (Subacute injury)
* Testosterone Deficiency defined as < 300ng/dL

Exclusion Criteria:

* Overt cardiovascular disease assessed by a) medical history, b) physical examination c) electrocardiogram
* Anaphylaxis to betadine, lidocaine, iodine
* Active infection at time of enrollment.
* Recent surgery (<1 month) at time of enrollment.
* History smoking tobacco (currently or in the past 12 months)
* History of more than low-risk history of alcohol consumption
* History of drug abuse
* History of use of cardiovascular-acting (i.e. statins, beta-blockers) therapeutics
* History of other health habits, medications, and supplements that could influence the outcome measures deemed by principal investigators and investigative team.

Ages: 18 Years to 89 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male sex
Study Population: Only male participants of all races and ethnic backgrounds aged 18-89 with a history of motor complete (AIS A/B) paraplegia (NLI T3 or Below). Time since injury <6 months at time of enrollment and diagnosed with normal and low T (Testosterone Deficiency defined as < 300ng/dL)
Sampling Method: Non-Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2025-07-15 (Actual); Primary Completion 2028-07-14 (Estimated); Study Completion 2028-07-14 (Estimated)

PRIMARY OUTCOMES:
Endothelium-dependent vasodilation | Measured at baseline (without acetylcholine) and immediately after each acetylcholine dose for 3-5 minutes.
  Total forearm blood flow with be measured by strain gauge venous plethysmography under baseline conditions and under pharmacological manipulation with acetylcholine at increasing concentrations (8, 16, 32ug/ml).
Endothelium-independent vasodilation | Measured at baseline (without sodium nitroprusside) and immediately after each sodium nitroprusside dose for 3-5 minutes.
  Total forearm blood flow with be measured by strain gauge venous plethysmography under baseline conditions and under pharmacological manipulation with sodium nitroprusside at increasing concentrations (1, 2, 4ug/ml).
Tissue plasminogen activator release | Measured at baseline and immediately after each isoproterenol and sodium nitroprusside dose for 3-5 minutes.
  Net endothelial release or uptake of t-PA and PAI-1 (both antigen and activity levels) at each dose of isoproterenol and sodium nitroprusside will be calculated as the product of the arteriovenous concentration gradient and the infused forearm plasma flow. Arteriovenous concentration gradients for both t-PA and PAI-1 antigen and activity for each subject (at each time point) will be determined by subtraction of the values measured in simultaneously collected venous and arterial blood samples
Endothelial cell-derived microvesicles concentration | Baseline
  Endothelial cell-derived microvesicles will be collected from venous blood samples and counted used flow cytometry to determine a circulating concentration.
Endothelial cell-derived microvesicles effects of human coronary artery endothelial cells nitric oxide bioavailability. | Baseline
  Endothelial cell-derived microvesicles will be sorted and collected by fluorescence-activated cell sorting (FACS) flow cytometry. The endothelial cell-derived microvesicles will be co-cultured with human coronary artery endothelial cells. Endothelial Nitric Oxide Synthase and phosphorylation sites of interest will be measured by intracellular protein expression quantification of whole cell lysates by capillary electrophoresis immunoassays. Nitric oxide production will be assessed by total nitric oxide and nitrate/nitrite parameter assays
Endothelial cell-derived microvesicles effects of human coronary artery endothelial cells reactive oxygen species and antioxidant capacity | Baseline
  Endothelial cell-derived microvesicles will be sorted and collected by fluorescence-activated cell sorting (FACS) flow cytometry. The endothelial cell-derived microvesicles will be co-cultured with human coronary artery endothelial cells. Super oxide dismutase and catalase expression will be measured by intracellular protein expression quantification of whole cell lysates by capillary electrophoresis immunoassays. Intracellular oxidative stress will be assessed by ROS-Glo H2O2 assay.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Park, MD, Principal Investigator — Craig Hospital
Locations (1):
- Craig Hospital, Englewood, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
Data sharing will be facilitated through active participation in Open Data Commons for SCI (ODC-SCI). ODC-SCI is a cloud-based community-governed repository to store, share, and publish research data on Spinal Cord Injury and is compliant with requirements for FAIR and trustworthy repositories established by NIH.